CLINICAL TRIAL: NCT03445234
Title: The Combined Influence of Blueberry and Banana Consumption on Metabolic Recovery From 75-km Cycling Exercise Stress
Brief Title: Blueberries, Bananas, Exercise Recovery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Appalachian State University (Other)
Collaborators: Dole Food Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 17-0352
Record Dates: First submitted 2017-08-10; First posted 2018-02-26 (Actual); Last update posted 2018-02-26 (Actual); Status verified 2018-01

CONDITIONS: Inflammatory Response; Metabolic Disturbance; Immune Suppression
Keywords: exercise; innate immune function; metabolomics; inflammation
MeSH Terms: conditions — Motor Activity; Inflammation | interventions — blueberry extract

STUDY DESIGN:
Intervention Model Description: Randomized parallel group
Who Masked: Participant, Investigator
Masking Description: Blueberry freeze dried powder or placebo powder
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Blueberry (Experimental): Freeze-dried blueberry powder
  Interventions: Dietary Supplement: Blueberry
- Placebo (Placebo Comparator): Placebo powder
  Interventions: Dietary Supplement: Placebo
- Banana (Experimental): Acute banana ingestion
  Interventions: Dietary Supplement: banana
- No banana (Experimental): No banana ingestion
  Interventions: Dietary Supplement: No banana

INTERVENTIONS:
Dietary Supplement: Blueberry — 26 g/day freeze-dried powder, 2 weeks duration
  Other Names: Placebo
  Arms: Blueberry
Dietary Supplement: Placebo — Placebo powder
  Arms: Placebo
Dietary Supplement: banana — Acute ingestion of bananas 0.2 g carb/kg every 15 min exercise with water
  Arms: Banana
Dietary Supplement: No banana — water only
  Arms: No banana

SUMMARY:
The PURPOSE of this study is to investigate the combined influence of 2-weeks blueberry ingestion and banana ingestion (during exercise) on performance and in mitigating metabolic perturbation, immune dysfunction, and increase in inflammation following a 75-km cycling time trial. We hypothesize that the combination of 2-weeks ingestion of blueberries (versus placebo) and acute ingestion of bananas (versus water alone) during 75-km cycling will:

1. Enhance performance.
2. Attenuate the magnitude of metabolic perturbation due to exercise (using a targeted panel of metabolites) which may be associated with increased plasma levels of beneficial gut-derived phenolics.
3. Attenuate post-exercise inflammation (as measured with cytokines, muscle damage markers, regulatory lipid mediators, ex-vivo monocyte cell cultures, and targeted immune proteins including S100A8 and S100A12).
4. Counter post-exercise downturns in innate immune function (natural killer cell lytic activity), and viral defense (using an ex-vivo cell culture with Hela cells).

DETAILED DESCRIPTION:
LAB VISIT #1: ORIENTATION AND BASELINE TESTING (about 1.5 hours):

One to two weeks prior to the start of the study, study participants will report to the NCRC Human Performance Lab for orientation and baseline testing. Study participants will be screened to verify "low risk" status for cardiovascular disease, and provide voluntary consent. Demographic and training histories will be acquired with questionnaires. Study participants will be tested for VO2max (i.e., maximal oxygen consumption) using the Lodi cycle ergometer. Percent body fat will be measured using the BodPod. Study participants will sit inside the BodPod with a tight-fitting swim suit for about 10 minutes while body fat is calculated.

LAB VISIT #2: START OF 2-WEEK SUPPLEMENTATION PERIOD (about 20 minutes)

On the assigned date and time, study participants will return to the lab in an overnight fasted state (9 or more hours with no food or beverage including coffee and tea, other than water). A blood sample will be collected from an arm or hand vein by trained phlebotomists. Each blood sample will not exceed 35 ml (2.3 tablespoons), and will be analyzed for indicators of immune function, inflammation, muscle damage, stress hormones, and indicators of plant polyphenol metabolism.

Study participants will be randomized to blueberry and placebo groups, and be given a 14-day supply of freeze-dried blueberry powder or placebo powder. The blueberry and placebo supplements will be ingested daily for 2-weeks prior to participation in the 75-km cycling time trial, the day of the exercise trial (after the blood draw, and supplied at the lab), and one day of recovery (after the blood draw, and supplied at the lab (thus 16 days total). The blueberry powder supplement (26 g per day or approximately one cup fresh blueberries equivalent) will consist of freeze-dried wild blueberries prepared by Future Ceuticals (Momence, IL). This product contains all of the polyphenols (in particular, anthocyanins), fiber, and natural sugars contained in fresh wild blueberries. The placebo powder will look identical but not contain freeze-dried blueberries. The placebo blueberry powder will consist of blueberry flavoring (2.8%), coloring (0.7% artificial purple, 0.3% artificial red), maltodextrin (21%), fructose (3.5%), citric acid (0.7%), and a silica flow agent (0.5%). Study participants will consume the blueberry and placebo powders by mixing them in fruit juices, yogurts, milk, or other products during the first meal of each day for two weeks. The blueberry and placebo powders should be stored in the freezer section of the refrigerator in the containers supplied to study participants.

LAB VISIT #3: POST-SUPPLEMENTATION LAB VISIT WITH 75-km CYCLING (about 8-9 hours)

* During the 3-day period prior to the 75-km cycling trial, study participants will taper exercise training and ingest a moderate-carbohydrate diet, with foods chosen from a food list moderating use of high fat foods, visible fats, and fruit/vegetable polyphenols. Study participants will record all food and beverage intake during the 3-day period.
* After the 2-week supplementation period, study participants will return to the lab at 7:00 am in an overnight fasted and rested state (on the same day of the week and time as the pre-supplementation lab visit).

  * Study participants will turn in the 3-day food record.
  * Study participants will verify that they have ingested the assigned supplement each day.
  * A 35 ml blood sample will be collected.
  * Study participants will next ingest 26 g of freeze-dried blueberry powder or placebo powder in 1.5 cups of water (with Equal packets available to improve taste as desired).
  * A simple questionnaire will be used for study participants to indicate muscle soreness (DOMS).
  * Study participants will complete a symptom log, which will include questions on digestive and mental health (heartburn, bloating, diarrhea, nausea, energy levels, ability to focus, etc.). Study participants will indicate responses using a 12-point Likert scale, with 1 relating to "none at all", 6 "moderate", and 12 "very high".
  * Study participants will be randomized to cycle 75-km on water alone or with bananas and water (and this will be revealed after the blood draw). Twenty minutes after ingesting the supplement, study participants will start the 75-km cycling time trial.

    75-km CYCLING TIME TRIAL

7:30 am: Start 75-km cycling time trial. Study participants are to complete the 75-km course as fast as possible.

* Study participants will use their own bicycles on CompuTrainer Pro Model 8001 trainers (RacerMate, Seattle, WA). A mountainous 75-km course with moderate difficulty will be utilized using the CompuTrainer software system.
* Heart rate and rating of perceived exertion (RPE) will be recorded every 30 minutes, and workload (watts) continuously monitored using the CompuTrainer MultiRider software system (version 3.0, RacerMate, Seattle, WA).
* Oxygen consumption, carbon dioxide production, and ventilation will be measured using the Cosmed metabolic cart after 16 km and 55 km cycling (through a facemask similar to what occurred during baseline testing). Performance will be monitored throughout the 75-km cycling time trial using percentage of maximal watts to ensure that a full effort is being given.
* Study participants will consume 3 ml/kg water every 15 min (e.g., about one cup for a 75 kg cyclist).
* If randomized to ingest bananas with water: Study participants will ingest Cavendish bananas, with the volume adjusted to 0.2 g carbohydrate/kg body weight every 15 minutes (or 0.8 g/kg carbohydrate per hour) during the 75-km time trials. For a 75-kg cyclist, fruit intake will be approximately one-half banana every 15 minutes. Bananas will be provided by Dole Foods at the appropriate ripening stage (full yellow, stage six). No other beverage or food containing energy or nutrients will be allowed during the cycling time trials.

  ~10:00-11:30 am: Immediate-post-exercise, 1.5-h recovery blood samples; lunch
* Blood samples will be taken from the arm vein immediately after completing the 75-km time trial, and then at 1.5-h post-exercise.
* Immediately post-exercise, study participants will complete the symptom log.
* Study participants will indicate muscle soreness using the DOMS questionnaire immediately post-exercise and 1.5-h post-exercise.
* Study participants will ingest no food or beverage other than water (7 ml/kg or about two cups during the 1.5 h post-exercise period).
* Right after the 1.5-h recovery blood sample has been collected, study participants will ingest a meal adjusted to 12 kcal/kg body weight. The meal will be prepared by Dole Foods and include grilled chicken, rice, corn, green beans, salt, and water.

  ~11:30 am to 3:00 pm: 3-h and 5-h recovery
* Additional blood samples and DOMS responses will be collected 3-h and 5-h post-exercise. During this time, study participants will rest quietly in the lab.

LAB VISITS #4 and #5: RECOVERY DAY BLOOD SAMPLES, 7:00 am:

• Study participants will return to the lab the following two mornings in an overnight fasted state at about 7:00 am (~21-h and 45-h after completing the 75-km time trial). Blood samples and responses to the DOMS questionnaire will be collected at both lab visits. Study participants will ingest the blueberry or placebo powder in the lab on the first recovery day following the blood sample collection.

ELIGIBILITY:
Inclusion Criteria:

* Male or female.
* Ages 18-55 years.
* Non-smoker.
* Regularly compete in road races (category 1 to 5) and/or are capable of cycling 75 km in a laboratory setting (using own bicycles on CompuTrainer training systems).
* Agree to train normally, maintain weight, and avoid the regular use of large-dose vitamin and mineral supplements, herbs, and medications that influence inflammation and immune function (especially Advil, Motrin, aspirin, and similar anti-inflammatory drugs) for the duration of the 2.5-week study. If in doubt, please discuss your supplement and medication use with the Research Manager during orientation (Courtney Goodman).
* Categorized as "low risk" using the American College of Sports Medicine screening questionnaire.
* Generally healthy and without chronic disease including cardiovascular disease (e.g., heart disease, stroke), cancer, type 1 and 2 diabetes, rheumatoid arthritis.

Exclusion Criteria:

* Inability to comply with study requirements.
* Body weight below 100 pounds.
* Pregnant or breastfeeding.
* Any other concurrent condition which, in the opinion of the primary investigator (PI), would preclude participation in this study or interfere with compliance.
* Current diagnosis of cardiovascular disease, diabetes, or cancer (except for non-melanoma skin cancer).
* History of allergic reactions to blueberries or bananas.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2017-09-11 (Actual); Primary Completion 2017-12-15 (Actual); Study Completion 2017-12-15 (Actual)

PRIMARY OUTCOMES:
Inflammation | Change from pre-supplementation to post-2-weeks supplementation, and to six post-exercise time points (0, 1.5, 3.0, 5.0, 21, 45 hours)
  Cytokines

SECONDARY OUTCOMES:
Metabolite shifts | Change from pre-supplementation to post-2-weeks supplementation, and to six post-exercise time points (0, 1.5, 3.0, 5.0, 21, 45 hours)
  Targeted panel of metabolites
Natural killer cell activity | Change from pre-supplementation to post-2-weeks supplementation, and to six post-exercise time points (0, 1.5, 3.0, 5.0, 21, 45 hours)
  Innate immune function
Exercise performance | After the 2-week period of blueberry or placebo intake
  75-km cycling time trial, with or without bananas
Targeted proteomics | Change from pre-supplementation to post-2-weeks supplementation, and to six post-exercise time points (0, 1.5, 3.0, 5.0, 21, 45 hours)
  Targeted panel of 24 immune proteins including S100A8 and S100A12
Muscle damage | Change from pre-supplementation to post-2-weeks supplementation, and to six post-exercise time points (0, 1.5, 3.0, 5.0, 21, 45 hours)
  Creatine kinase
Lipid mediators | Change from pre-supplementation to post-2-weeks supplementation, and to six post-exercise time points (0, 1.5, 3.0, 5.0, 21, 45 hours)
  Arachadonic acid oxidized derivatives from LC-MS-MS analysis

CONTACTS AND LOCATIONS:
Overall Officials: David C. Nieman, DrPH, Principal Investigator — Appalachian State Univ
Locations (1):
- North Carolina Research Campus, Human Performance Lab, Kannapolis, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No